CLINICAL TRIAL: NCT04262024
Title: Clinical Guidance to Increase Women's Awareness of Some Contributing Factors to Help Proper Treatment of Unexplained Resistant Hyperprolactinemia Not Responding to Therapeutic Dopamine Agonists (DA)
Brief Title: Clinical Guidance for Proper Treatment of Unexplained Resistant Hyperprolactinemia.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Professor Atef Darwish, Professor of Obstetrics and Gynecology, Woman's Health University Hospital, Egypt
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: Clinical trial
Record Dates: First submitted 2020-02-01; First posted 2020-02-10 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Health Education
Keywords: health education; prolactin; hyperprolactinemia; resistant
MeSH Terms: conditions — Health Education; Hyperprolactinemia | interventions — Cabergoline

STUDY DESIGN:
Intervention Model Description: Prospective study ( randomized controlled trial)
Who Masked: Participant
Masking Description: Hyperprolactinemic women receiving cabergoline therapy will be divided into 2 groups: with health education and without health education.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Women with hyperprolactinemia are scheduled for cabergoline therapy cabergoline 1.5-2 mg/week. for one month plus health education.
  Interventions: Drug: cabergoline 1.5-2 mg/week).orally daily for 1 month plus health education
- Group B (Active Comparator): Women with hyperprolactinemia are scheduled for cabergoline therapy 1.5-2 mg/week. for one month without health education.
  Interventions: Drug: cabergoline 1.5-2 mg/week).orally daily for 1 month without health education

INTERVENTIONS:
Drug: cabergoline 1.5-2 mg/week).orally daily for 1 month plus health education — Women with hyperprolactiemia scheduled for cabergoline therapy 1.5-2 mg/week). for one month will be offered health education to help minimize prolactin level(group A)
  Other Names: cabergoline 1.5-2 mg/week+health education
  Arms: Group A
Drug: cabergoline 1.5-2 mg/week).orally daily for 1 month without health education — Women with hyperprolactiemia scheduled for cabergoline 1.5-2 mg/week).for one month will not be offered health education (group B)
  Other Names: cabergoline 1.5-2 mg/week
  Arms: Group B

SUMMARY:
Many women despite being well-treated in proper dose, with proper drug and for proper duration, may not respond to different forms of prolactin normalizing drugs.

This will lead to extension of the treatment duration up to months or even years.

Doctors usually increase the dose of the drug with high possibility of side effects and even complications. Some doctors change drug group to another without any significant improvement of hyperprolactinemia. hyperprolactinemia can indicate a deeper issue, about 10 percent of the population has hyperprolactinemia. Life style, feeding habits and sexual behaviors are usually not included in the management protocols of hyperprolactinemia.

Aim of the study:

This study will be aimed to:

test the impact of clinical guidance to increase women's awareness of some contributing factors to help proper treatment of unexplained resistant hyperprolactinemia not responding to therapeutic DA (cabergoline 1.5-2 mg/week).

Hypothesis of the study:

H1- Health education for women under drugs of hyperprolactinemia is effective to reduce the level of prolactin.

H0- Health education for women under drugs of hyperprolactinemia is not effective in reducing the level of prolactin

DETAILED DESCRIPTION:
Subjects and methods:

All women diagnosed to have hyperprolactinemia as diagnosed by one laboratory (lab of the Woman's Health University Hospital).

Research Design:

Prospective study (randomized controlled trial) .

Setting:

This study will be conducted at the outpatient clinic of the Woman's Health University Hospital, Assiut University.

Sample size: convenience sample started from February 2020 to January 2023 or reached 120 cases, 60 in each arm.

Statistical analysis

Data entry and statistical analysis will be done using the statistical package for social science program (SPSS. version 22). Qualitative variables will be presented as number and percentage. Quantitative variables will be presented as mean +SD. Comparison between qualitative variables will be done by using chi-square. Comparison between quantitative variables will be done by using student t-test.

ELIGIBILITY:
Inclusion criteria:

1. Pathologic hyperprolactinemia due to any cause.
2. Non-pregnant.
3. Not lactating.

Exclusion criteria:

1. Physiologic hyperprolactinemia.
2. Women who don't consent for follow up.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Achievement of normoprolactinemia after one month of therapy of hyperprolactinemia | 1 month
  response of hyperprolactinemic women to carbergoline o.5 mg for one month with or without health education by a nurse to achieve normoprolactinemia.

CONTACTS AND LOCATIONS:
Overall Officials: Atef M Darwish, Prof, Principal Investigator — Prof.
Locations (1):
- Woman's Health University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No